CLINICAL TRIAL: NCT03543774
Title: Lipid-lowering Regimes Improve Oxidative Stress, Tryptophan Degradation in Hypercholesterolemia Chronic Kidney Disease Patients
Brief Title: Lipid-lowering Therapies in Vietnamese Chronic Kidney Disease Population
Acronym: VietCKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hue University of Medicine and Pharmacy (Other)
Collaborators: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Duong Thi Ngoc Lan, Principal Investigator, Physician, Master degree, Hue University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HueUMP
Record Dates: First submitted 2018-04-17; First posted 2018-06-01 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Hypercholesterolemia; Chronic Kidney Diseases
Keywords: Chronic kidney disease; Lipid lowering therapy; Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Renal Insufficiency, Chronic | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- simvastatin treatment (Active Comparator)
  Interventions: Drug: Simvastatin 40mg
- EZE/simvastatin 10/20 mg treatment (Sham Comparator)
  Interventions: Drug: Ezetimibe/simvastatin 10/20 mg/day
- EZE/simvastatin 10/40 mg treatment (Sham Comparator)
  Interventions: Drug: Ezetimibe/simvastatin 10/40 mg/day

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin mono-therapy at the dose of 40 mg/day for 12 months
  Arms: simvastatin treatment
Drug: Ezetimibe/simvastatin 10/20 mg/day — Ezetimibe/simvastatin combined therapy at the dose of 10/20 mg/day for 12 months
  Arms: EZE/simvastatin 10/20 mg treatment
Drug: Ezetimibe/simvastatin 10/40 mg/day — Ezetimibe/simvastatin combined therapy at the dose of 10/40 mg/day for 12 months
  Arms: EZE/simvastatin 10/40 mg treatment

SUMMARY:
This study aims to determine the mechanisms underlying dyslipidemia in chronic kidney disease (CKD) and effect of lipid-lowering therapies in patients with CKD via parameters of lipid, oxidative stress, tryptophan delegation as well as renal function and side effects. Thirty 3,4 CKD patients with low-density lipoprotein (LDL) > 100 mg/mL (2,59mmol/l), randomly receive three different LDL lipid-lowering therapies: Simvastatin (40 mg/day) or ezetimibe/simvastatin combination (10/20 mg/day or 10/40 mg/day).

DETAILED DESCRIPTION:
The prevalence of chronic kidney disease (CKD) in Vietnamese population is increasing along with hypertension and diabetes. In CKD patient, cardiovascular disease (CVD) is the leading cause of mortality. The lipidemic disorder is one of the CV risk factors in CKD but it was not fully concerned in Viet Nam.

Hypocholesterolemia therapy has shown many benefits; however, its effects on OS and endothelial function are still not fully evidenced.

In clinical practice, physicians always concern the effects and safety before giving the prescription. However, despite the high frequency of statin treatment, only 1/3 of CKD patients achieved the LDL-C goal. Whether high-dose of statins mono-therapy is more effective in LDL-C lowering is still unclear, but are associated with a high rate of hepatotoxicity, myopathy.

Lowering LDL-C with statin mono-therapy and statin/ezetimibe combination reduces the risk of CVD in population without kidney disease. Which Cholesterol-lowering therapies are suitable for stage 3,4 CKD patients in term of e-GFR reduction and side effects? There is no data related to this field in the Vietnamese CKD population.

Thus, more advanced lipid-lowering therapies and a better understanding of the mechanism is needed for treatment strategy of hyperlipidemia in Vietnamese patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study:

  * ≥ 50 years old but not treated with chronic dialysis or kidney transplantation
  * In adults aged 18-49 years with CKD but not treated with chronic dialysis or kidney transplantation, statin treatment in people with one or more of the following: known coronary disease (myocardial infarction or coronary revascularization); diabetes mellitus; prior ischemic stroke; estimated 10-year incidence of coronary death or non-fatal myocardial infarction > 10%.
* CKD in the 3,4 stage: (e-GFR: 15-60 ml/min/1.73 m2)
* CKD proteinuria (defined as Creatinine clearance >20 ml/min/1.73 m2 combines with urinary protein excretion rate >300mg/24 h)
* LDL cholesterol concentration > 100 mg/dl (2,59 mmol/l)

Exclusion Criteria:

In adults with dialysis-dependent CKD

* Heart failure (New York Heart Association class III or more)
* Previous or concomitant treatment with corticoids, statin, immunosuppressive agents, vitamin B6, B12, folate.
* Pregnancy
* Patients who do not agree to participate the research
* Patients are unable to understand the purposes and the risks of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
To measure the serum level of TC, LDL-C, HDL-C, TG, Creatinine, uric acid, and allantoin in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The serum level of TC, LDL-C, HDL-C, TG, Creatinine, uric acid, and allantoin will be measured in mg/dL.
To measure the serum level of Taurine, Tryp, and Kyn in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The serum level of Taurine, Tryp, and Kyn will be measured in micromol/L
To measure the number of red blood cell, white blood cell and platelet in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The number of red blood cell, white blood cell, and platelet will be measured in number/L
To measure the serum level of MDA in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The serum level of MDA will be measured in nmol/L
To measure the level of Albuminuria and urine Creatinine in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The serum level of Albuminuria and urine Creatinine will be measured in mg/dL
To measure the serum level of SGOT, SGPT, and Creatinin Kinase in Vietnamese CKD population and in healthy persons at the base time. | At the base time
  The serum level of SGOT, SGPT and Creatinin Kinase will be measured in Units/L

SECONDARY OUTCOMES:
To measure the serum level of TC, LDL-C, HDL-C, TG, Creatinine, uric acid, and allantoin in Vietnamese CKD population at 4th, 8th, 12th month. | at 4th, 8th and 12th month
  The serum level of TC, LDL-C, HDL-C, TG, Creatinine, uric acid, and allantoin will be measured in mg/dL.
  The change of results during treatment will be described and will be compared in 3 different groups
To measure the serum level of Taurine, Tryp, and Kyn in Vietnamese CKD population at 4th, 8th, 12th month. | at 4th, 8th and 12th month
  The level of Taurine, Tryp, and Kyn will be measured in micromol/L. The change of results during treatment will be described and will be compared in 3 different groups
To measure the number of red blood cell, white blood cell and platelet in Vietnamese CKD population at 4th, 8th, 12th month. | at 4th, 8th and 12th month
  The number of red blood cell, white blood cell, and platelet will be measured in number/L.
  The change of results during treatment will be described and will be compared in 3 different groups
To measure the serum level of MDA in Vietnamese CKD population at 4th, 8th, 12th month. | at 4th, 8th and 12th month
  The serum level of MDA will be serum in nmol/L. The change of results during treatment will be described and will be compared in 3 different groups
To measure the serum levels of SGOT, SGPT and Creatinine Kinase in Vietnamese CKD population at 4th month, 8th month and the 12th month | at 4th, 8th and 12th month
  The unexpected effects of each treatment therapy on the liver and on the muscle will be accessed by measuring the level of SGOT, SGPT and Creatinine Kinase. These laboratory test will be measured at 4th month, 8th month and the 12th month. These results will be compared in 3 different groups
To measure the level of Albuminuria and urine Creatinine in Vietnamese CKD population at 4th, 8th, 12th month. | at 4th, 8th and 12th month
  The level of Albuminuria and urine Creatinine will be measured in mg/dL. The change of results during treatment will be described and will be compared in 3 different groups

CONTACTS AND LOCATIONS:
Overall Officials: Duong Thi Ngoc Lan, Master, Principal Investigator — Hue University of Medicine and Pharmacy
Locations (1):
- Hue University of Medicine and Pharmacy, Huế, Thừa Thiên Huế Province, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- See also: A Trial of Pitavastatin Versus Rosuvastatin for Dyslipidemia in Chronic Kidney Disease — https://www.jstage.jst.go.jp/article/jat/22/12/22_29264/_pdf/-char/en
- See also: Effects of lowering LDL cholesterol on progression of kidney disease — http://jasn.asnjournals.org/content/25/8/1825.long
- See also: Ezetimibe and simvastatin for the prevention of cardiovascular events in predialysis chronic kidney disease patients: a review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3534534/
- See also: The effects of lowering LDL cholesterol with simvastatin plus ezetimibe in patients with chronic kidney disease (Study of Heart and Renal Protection): a randomised placebo-controlled trial. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3145073/

DOCUMENTS (3):
  • Study Protocol (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03543774/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT03543774/SAP_001.pdf
  • Informed Consent Form (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03543774/ICF_002.pdf